CLINICAL TRIAL: NCT05138107
Title: Prospective Placebo-controlled Study of Synochi Scar Spray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Synochi, LLC (Industry)
Collaborators: LAC+USC Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SYNSS_02
Record Dates: First submitted 2021-11-09; First posted 2021-11-30 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Burns Multiple
Keywords: autologous skin transplant; appearance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Graft Burn Patients Experimental Site (Experimental): Both placebo and active cosmetic scar spray will be applied to different parts of the same scar on each participant. The active and the placebo spray will both be applied to the designated area of each scar twice per day. The amount sprayed will cover the designated area of the scar and then be massaged into to scar and surrounding skin with each application. This will be done twice daily for the nine-month duration of the study.
  Interventions: Other: Synochi Scar Spray Cosmetic
- Skin Graft Burn Patients Placebo Site (Placebo Comparator): Both placebo and active cosmetic scar spray will be applied to different parts of the same scar on each participant. The active and the placebo spray will both be applied to the designated area of each scar twice per day. The amount sprayed will cover the designated area of the scar and then be massaged into to scar and surrounding skin with each application. This will be done twice daily for the nine-month duration of the study.
  Interventions: Other: Synochi Scar Spray Placebo

INTERVENTIONS:
Other: Synochi Scar Spray Cosmetic — Application of the cosmetic on each skin graft in a blinded fashion in different sections for a 9 month duration.
  Arms: Skin Graft Burn Patients Experimental Site
Other: Synochi Scar Spray Placebo — Application of the placebo on each skin graft in a blinded fashion in different sections for a 9 month duration.
  Arms: Skin Graft Burn Patients Placebo Site

SUMMARY:
Randomized, double-blind, placebo controlled, prospective, split-scar study of severe burn victims with autologous skin transplants. 9 months intervention time and 3 months follow-up, photographic scar documentation, self-and observer questionnaires throughout

DETAILED DESCRIPTION:
Interventional, comparative, prospective, evaluator blinded, randomized, placebo- controlled, split-scar model longitudinal study including 28-31 healthy study participants (See Section 6 Statistical Considerations) with both the original burn scar area that is the skin graft recipient area and the skin graft donor site.

ELIGIBILITY:
Inclusion Criteria:

* - Study participants are healthy study participants from any sex and race, but must be between 22 and 50 years of age at the time of consent.
* Study participants must be willing to provide written informed consent and be able to read, write, speak, and understand the test procedures in English. Ability will be documented with a doctors' note.
* Study participants must be willing to sign a Photo and Video Release Form.
* Study participants must possess both the original burn scar area that is the skin graft recipient area and the skin graft donor site that is at least around 6 weeks old that have not been altered in any way prior (No prior scar reduction surgery, laser, steroid injections, silicone sheets or anything of the like).
* Study participants must be in good general health.

Exclusion Criteria:

* - Study participants must not currently be under the care of a medical or cosmetic professional for care of the scar to be evaluated in testing.
* They must be without medical diagnosis of medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an organ transplant, a heart murmur, mitral valve prolapse with heart murmur, fibromyalgia, ulcerative colitis, Crohn's disease, moderate to severe asthma (requiring daily use of systemic steroid medication, nasal steroids are permitted), an immunocompromised condition such as AIDS (or HIV positive), lupus, or medicated multiple sclerosis, not pregnant or trying to become pregnant, lactating, transplant recipient on immunosuppression, the BMI should be 19 - < 35.
* Have any type of vascular disease (e.g., arteriosclerosis, Raynaud's Syndrome, or peripheral venous disease) or any blood clotting disorders.
* Have participated in another clinical study within the past 14 days, or be currently participating in another clinical study.
* Have or have someone in their household with known sensitivities or allergies to latex (rubber), bar or liquid cleansing products, serums, moisturizers, lotions, creams, preservatives, fragrances, cosmetics, or common ingredients used in traditional Chinese medicine, including Notopterygium root (Notopterygium Incisum), sweetgum fruit ( Liquidambaris Fructus), bur reed rhizome (Rhizoma Sparganii), corydalis rhizome (Rhizoma Corydalis), ledebouriella root / siler (Radix Saposhnikoviae), costus root (Radix Auklandiae Lappae), rehmannia root (Radix Rehmanniae Preparata), deer horn gelatin/glue (Gelatinum Cornu Cervi), safflower (Carthamus Tinctorius), forsythia fruit (Fructus Forsythiae), red earthworm (Lumbricus), trichosanthes root (Radix Trichosanthes), Chinese motherwort (Herba Leonuri), millettia vine (Caulis Spatholobi), zedoary rhizome (Rhizoma Curcumae), turmeric tuber (Radix Curcumae), rhubarb (Radix et Rhizoma Rhei), white peony root (Radix Paeoniae Alba), white mustard seed (Semen Sinapis Albae), Chinese angelica root (Angelicae sinensis Radix), cinnamon twig (Ramulus Cinnamomi), red peony (Radix Paeoniae Rubra), peach kernel (Semen Persicae), astragalus (Radix Astragali), frankincense resin (Resina Boswelliae Carterii), myrrh (Resina Commiphorae Myrrhae), sandalwood (Santalum Album), radiz notoginseng (Radix Notoginseng), spine of honey locust (Spina Gleditsiae), silkworm (Bombyx Batryticatus)
* Have experienced hives (raised welts) as a reaction to anything contacting their skin.
* Not be diagnosed with a medical condition that, in the opinion of the Principal Investigator, would preclude participation.
* Not be unwilling to fulfill the performance requirements of the study.
* Not be direct employees, in a relationship with, or family of the sponsor or Principal Investigator.
* Not be participating in any other clinical trial during the time of this clinical trial.
* Medication: Not be receiving any steroid medications (including those used to treat asthma) other than for contraception, hormone therapy, or menopausal purposes. No chemotherapeutic agents or any medication that interferes with wound healing (rheumatologic agents, Emgality or Aimovig).

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-05-17 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
improvement of cosmetic appearance Synochi Scar Spray versus Placebo | 12 month study time frame
  Section I of the Patient Scar Assessment Questionnaire (9 questions) minimum 9 points, maximum 36 with higher ratings indicating less improvement of cosmetic appearance

SECONDARY OUTCOMES:
evaluate the safety of Synochi Scar Spray | 12 month study time frame
  Safety of Synochi Scar Spray as indicated by absence of adverse events and/or severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gillenwater, MD, Principal Investigator — USC School of Medicine

IPD SHARING:
Plan to Share IPD: No